CLINICAL TRIAL: NCT07063875
Title: Supplementing With IL-2 to Verifiably eRadicate Radiological Progression
Brief Title: Adding IL-2 to Tebentafusp to Eradicate Cancer Progression
Acronym: SILVER
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: St Vincent's Hospital, Sydney (Other)
Responsible Party: Principal Investigator, Anthony Joshua, FRACP, Professor, St Vincent's Hospital, Sydney
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SILVER Trial
Record Dates: First submitted 2025-06-17; First posted 2025-07-14 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Uveal Melanoma; Metastatic Uveal Melanoma; Metastatic Uveal Melanoma in the Liver
Keywords: metastatic uveal melanoma; Immunotherapy; Treatment resistance; Combinational immunotherapy
MeSH Terms: conditions — Uveal Melanoma | interventions — aldesleukin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment arm (Experimental): Single arm study -all enrolled participants will receive investigational products- IL-2 (Proleukin) and Tebetafusp
  Interventions: Drug: Aldesleukin

INTERVENTIONS:
Drug: Aldesleukin — IL-2 in combination with Tebentafusp
  Other Names: Proleukin

SUMMARY:
A recent clinical trial found that after 36 months, patients taking tebentafusp had a median survival of 21.6 months, compared to 16.9 months for those in the control group. Since recruitment for tebentafusp in metastatic uveal melanoma (mUM) has ended, a new trial is starting to test whether adding IL-2 can help overcome resistance to tebentafusp and improve its effectiveness.

This study aims to answer:

1. Can combining tebentafusp with IL-2 improve tumor response and overall survival?
2. What are the benefits and side effects of this combination therapy?

All participants will receive both IL-2 and tebentafusp in a 28-day treatment cycle. The dosing schedule is as follows:

Cycle1:

Day1-3 IL-2 Day4 Tebentafusp Day 10 IL-2 Day 11 Tebentafusp Day 17 IL-2 Day 18 Tebentafusp Day 24 IL-2 Day 25 Tebentafusp

Cycle 2 & thereafter Day 1 IL-2 Day 2 Tebentafusp Day 8 IL-2 Day 9 Tebentafusp Day 15 IL-2 Day 16 Tebentafusp Day 22 IL-2 Day 23 Tebentafusp

DETAILED DESCRIPTION:
Uveal melanoma (UM) is a rare and highly malignant neoplasm affecting the vascular layers of the eye (iris, ciliary body, or choroid). UM primarily metastasizes to the liver and less commonly to the lungs and bones. Once patients develop mUM, the prognosis is very poor with a median survival of < 12 months. There are limited treatments for mUM that extend survival, and there is no proven standard of care. Enrolment in investigational clinical trials is the treatment option recommended by national and regional guidelines. A clear unmet medical need exists for patients with this serious and life- threatening disease.

Tebentafusp is a bispecific protein therapeutic comprising a soluble, affinity-enhanced T cell receptor (TCR; targeting domain) fused to an antibody single-chain variable fragment (scFv) targeting cluster of differentiation (CD)3 (effector domain). Tebentafusp recognizes a peptide derived from gp100, a melanocyte lineage antigen expressed strongly in tumors derived from melanocytes that is presented on the cell surface by HLA-A*02:01. Once the soluble TCR of tebentafusp is engaged, the scFv effector domain can bind to CD3 on any T cell, redirecting the T cell to produce effector cytokines and kill the cell presenting the target peptide. In addition, tebentafusp-mediated lysis may prime an endogenous antitumor immune response via epitope spreading. This mechanism is distinct from all other therapies that have been studied for melanoma.

The most recent evidence for the utility of Tebentafusp was just published demonstrating that at a minimum follow-up of 36 months, median overall survival was 21.6 months in the tebentafusp group and 16.9 months in the control group (hazard ratio for death, 0.68; 95% confidence interval, 0.54 to 0.87).

Now that all registrational metastatic trials in UM with Tebentafusp are closed to recruitment, this trial is being initiated to explore the addition of IL2 to offer a mechanism to overcome tebentafusp resistance and explore its efficacy and toxicities.

This Phase Ib study aims to administer tebentafusp in combination with IL-2 to improve primary endpoint of radiographic response rate as well the secondary endpoint of Overall Survival (OS).

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed metastatic UM or unresectable UM patients
2. HLA-A*02:01 positive
3. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1
4. RECIST 1.1 defined progression on single-agent Tebentafusp, with no other intervening systemic therapies

Exclusion Criteria:

1. Presence of untreated or symptomatic central nervous system (CNS) metastases, leptomeningeal disease, or cord compression. (NOTE: Participants with treated CNS lesions may enroll provided all of the following apply: Treated CNS lesions must be radiographically stable for ≥ 4 weeks after intervention (surgery and/or radiation). Participants must be neurologically stable off systemic corticosteroids for at least 2 weeks prior to trial entry, AND Greater than 14 days elapsed between the last dose of previous Tebentafusp and first dose of IL-2 on trial)
2. Systemic treatment with steroids or any other immunosuppressive drug use within 2 weeks of the planned first dose of program intervention, with the following exceptions: Treatment for well-controlled and asymptomatic adrenal insufficiency is permitted, but replacement dosing is limited to prednisone ≤ 10 mg daily or the equivalent; Local steroid therapies (eg, optic, ophthalmic, intra- articular, or inhaled medications) are acceptable.
3. Any relevant medical condition, which in the opinion of the treating physician, would prevent the participant enrolling into the Program due to concerns related to safety, compliance with procedures, or interpretation of program results.
4. Chronic viral infections as indicated below. NOTE: Testing for human immunodeficiency virus (HIV), hepatitis B virus (HBV), and hepatitis C virus (HCV) status prior to enrollment is not necessary unless clinically indicated.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Safety of Combination therapy | Through study completion, approx 1 year
  As assessed by CTCAE V5.0

SECONDARY OUTCOMES:
Radiological progression free survival | Through study completion, approx 1 year
  Time to RECIST 1.1 progression
Overall Survival | Through study completion, approx 1 year
  Time to Death

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Joshua, FRACP, Principal Investigator — St Vincent's Hospital, Sydney
Locations (2):
- Australia (2):
  - Kinghorn Cancer Centre, St. Vincent's Hospital, Sydney, New South Wales
  - Alfred Hospital, Melbourne, Victoria

IPD SHARING:
Plan to Share IPD: No